CLINICAL TRIAL: NCT01503879
Title: Effects of General Anaesthesia and Invasive Mechanical Ventilation on Alveolo-capillary Membrane: Evaluation of Gas Exchange by the Measurement of Lung Diffusion for Carbon Monoxide (DLCO) and Plasma Dosage of Surfactant Protein-B (SPB).
Brief Title: Evaluation of Gas Exchange by the Measurement of Lung Diffusion for Carbon Monoxide During General Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Prof. Roberto Fumagalli's, MD, San Gerardo Hospital
Other Study IDs: ARHSG 10 2010 DLCO1
Record Dates: First submitted 2011-12-31; First posted 2012-01-04 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Lung Diffusion; Acute Respiratory Failure
Keywords: general anaesthesia; invasive mechanical ventilation; DLCO; SPB

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — surfactant protein B
Oversight: Data Monitoring Committee: No

SUMMARY:
Mechanical ventilation is a therapeutic method used in order to keep gas exchange adequate to cell metabolism in patients with acute respiratory failure. It is currently proved that, although on one hand the use of this method keeps gas exchange, on the other hand it promotes and supports pulmonary inflammatory processes (VILI). A recent study about the effect of positive end-expiratory pressure (PEEP) on DLCO (diffusing capacity of the lung for carbon monoxide) in patients undergoing invasive mechanical ventilation has proved that patients without any evident pulmonary disease (negative medical history, negative chest clinical examination, normal chest X-ray radiography and normal arterial oxygen tension [PaO2]) after 24 hours of invasive mechanical ventilation show a significant worsening of pulmonary gas exchange properties. The authors have supposed that this worsening may be caused by an early alteration of alveolar-capillary membrane caused by mechanical ventilation itself. This hypothesis finds support in some studies carried out on animal models which founds that mechanical ventilation, even when low tidal volumes (Vt) are set for a few hours, is able to induce lung injury (as shown by histologic findings). The most sensitive and specific tools the investigators can currently rely on for the study of alveolar-capillary membrane are the measurement of diffusing capacity of the lung for carbon monoxide (DLCO) and the evaluation of plasmatic levels of pulmonary surfactant protein B (SPB). DLCO is a standard, widely diffused technique for the evaluation of functional alterations of alveolar-capillary membrane and it is currently available also for patients undergoing invasive mechanical ventilation. SBP is produced by type II pneumocytes in the alveoli. An increase of its plasmatic levels is correlated to a decay of pulmonary gas exchange; SPB thus can be considered an alveolar-capillary membrane anatomical damage marker.

The primary end-point of this study is to evaluate the changes of anatomical (SPB) and functional (DLCO) features of alveolar-capillary membrane between the spontaneous breathing and mechanical ventilation as well as the progressive changes affecting DLCO and SPB over time during general anaesthesia and mechanical ventilation in patients with otherwise healthy lung undergoing elective surgery. This in order to check the timing of the observed worsening of alveolar-capillary membrane function, and to find out if the process is progressive in time.

The secondary end point is to check if the alterations of functional features of alveolar membrane (DLCO) are proportionate to the increase of alveolar injury marker (SPB), in order to understand if the worsening of alveolar-capillary membrane function is to be attributable to an anatomical damage or to a physiologic change of the ventilation-perfusion matching.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* undergoing a non-thoracic, non-laparoscopic surgery, lasting more than three hours and requiring general anaesthesia and invasive mechanical ventilation

Exclusion Criteria:

* COPD 3 Gold stage or above
* ASA physical status classification system 4 or above
* heart failure NYHA 2 or above
* chronic kidney disease
* axillary temperature over 38 °C
* BMI over 30 kg/m^2
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery lasting more than three hours, requiring general anaesthesia and invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto MD Fumagalli, Principal Investigator — Milano Bicocca University
Locations (1):
- Ospedale San Gerardo, Monza, MB, Italy